CLINICAL TRIAL: NCT04046822
Title: Could Gut Microbiome Contribute to the Therapeutic Effect of Liraglutide 3.0 mg? A Randomized Double Blind Placebo Controlled Trial
Brief Title: Effect of Liraglutide on Microbiome in Obesity
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Annamaria Colao, Principal Investigator, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Microbiome 1
Record Dates: First submitted 2019-07-08; First posted 2019-08-06 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Obesity; Weight Loss; Microbiome
Keywords: obesity; liraglutide; gut microbiome
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Liraglutide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active drug (Active Comparator): Liraglutide is administered once daily by subcutaneous injections with the pen-injector, either in the abdomen, thigh or upper arm. Injections can be done at any time of day irrespective of meals. Subjects will be instructed to escalate the liraglutide dose to 3.0 mg/day over a 4 week period following an initial dose of 0.6 mg/day and weekly dose escalation steps of 0.6 mg/day.
  Interventions: Drug: Liraglutide 6 MG/ML [Saxenda]
- Placebo (Placebo Comparator): Placebo is administered once daily by subcutaneous injections with the pen-injector, either in the abdomen, thigh or upper arm. Injections can be done at any time of day irrespective of meals. Subjects will be instructed to escalate the placebo dose to 3.0 mg/day over a 4 week period following an initial dose of 0.6 mg/day and weekly dose escalation steps of 0.6 mg/day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide 6 MG/ML [Saxenda] — Liraglutide is administered once daily by subcutaneous injections with the pen-injector, either in the abdomen, thigh or upper arm. Injections can be done at any time of day irrespective of meals. Subjects will be instructed to escalate the liraglutide dose to 3.0 mg/day over a 4 week period following an initial dose of 0.6 mg/day and weekly dose escalation steps of 0.6 mg/day.
  Other Names: Saxenda
  Arms: Active drug
Drug: Placebo — Placebo is administered once daily by subcutaneous injections with the pen-injector, either in the abdomen, thigh or upper arm. Injections can be done at any time of day irrespective of meals. Subjects will be instructed to escalate the placebo dose to 3.0 mg/day over a 4 week period following an initial dose of 0.6 mg/day and weekly dose escalation steps of 0.6 mg/day.
  Other Names: Saline Injection
  Arms: Placebo

SUMMARY:
The purpose of the trial is to assess whether the beneficial effect of liraglutide on weight is mediated by changes in the composition of the intestinal Microbiome. The main mechanisms of action of liraglutide were traced to a reduction in the secretion of glucagon and slowing gastric emptying resulting in decreased appetite and body weight. It also seems that liraglutide is capable of increasing the satiety signals thanks to a dual mechanism of stimulation and inhibition induced by medication. Pomc neurons (opiomelacortin) present in hypothalamic arcuate nuclei, stimulated by liraglutide, glucagon-like peptide- 1 (GLP-1) receptor expressed by inhibiting intensely appetite. At the same time through the GABAergic neuronal activity is inhibited neuropeptide Y(NPY) deputies to the production of orexins that are powerful promoters of appetite. Alterations in the composition of the human gut microbiome occur in metabolic disorders such as obesity, diabetes. Liraglutide has been reported to switch microbiome composition towards lean-related bacterial phylotypes in animal studies. This leads to hypothesize that the switch of microbiome by liraglutide may be one of the mechanisms through which liraglutide may exert its effect. In particular the investigators hypothesize that liraglutide could restore a healthy microbiome or at least improve the microbiome composition through slowing gastrointestinal motility. Moreover, the liraglutide-related change of microbiome could be an additional mechanism that contribute to the beneficial metabolic effect of liraglutide. To test this hypothesis the investigators will investigate if there will be any change of gut microbiome assessed as Firmicutes-to-Bacteroidetes ratio after liraglutide treatment. In order to understand if the change of gut microbiome after liraglutide treatment occurs as an association or contributes to the effect of liraglutide ,the investigators will correlate the Firmicutes-to-Bacteroidetes ratios with the changes of Body Mass Index, Body Composition, appetite parameters, chronic inflammation parameters, lipid profile and insulin resistance. All the subjects will follow the same diet in order to avoid any bias.

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel group, placebo-controlled trial comparing liraglutide 3.0 mg with placebo both administered subcutaneously once-daily in subjects with established obesity. Subjects will be randomised in a 1:1 ratio to receive either liraglutide 3.0 mg or placebo as an adjunct to standard-of-care.All baseline assessments will be done prior to administration of the first dose of trial product while all the follow up assessments will be done at the end of the trial. Dose escalation of liraglutide/placebo will take place during the first 4 weeks after randomisation as described. All subjects will aim at reaching the recommended target dose of 3.0 mg liraglutide once-daily or the corresponding volume of placebo. In this trial approximately 70 subjects will be randomly assigned to trial product.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial;
2. Age ≥ 18 years and < 65 years at the time of signing informed consent;
3. Body mass index (BMI) ≥ 30 kg/m2
4. Stable body weight during the previous 3 months (< 5 kg self-reported weight change).

Exclusion Criteria:

General Safety

1. Current or history of treatment with medications that may cause significant weight gain for at least 3 months before this trial;
2. Current use or use within three months before this trial of GLP-1 receptor agonist, pramlintide, sibutramine, orlistat, zonisamide, topiramate or phentermine;
3. Type 1 diabetes;
4. Type 2 diabetes;
5. Obesity related to endocrine diseases;
6. Hepatic Failure (AST and/or ALT >3 times upper limit of normal and/or Total Bilirubin >1.7 upper limit of normal)
7. End stage renal disease (eGFR < 30 ml/min/1.73 m2 ) or chronic or intermittent haemodialysis or peritoneal dialysis
8. History or presence of chronic pancreatitis
9. Presence of acute pancreatitis within the past 180 days prior to the day of screening
10. Personal or first degree relative(s) history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma
11. Presence or history of malignant neoplasms within the past 5 years prior to the day of screening
12. Severe psychiatric disorder which in the investigator's opinion could compromise compliance with the protocol
13. Known or suspected hypersensitivity to trial product(s) or related products
14. Previous participation in this trial. Participation is defined as randomisation
15. Receipt of any investigational medicinal product within 30 days before screening
16. Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using a highly effective contraceptive method i.e.:

    * patients who use combined hormonal contraceptives (containing estreogen and progesterone) associated with inhibition of ovulation or oral, intravaginal that transdermal;
    * patients who use hormonal contraceptives based only progesterone that inhibit ovulation, whether oral, injectable or implantable
    * patients with placement of IUD (intrauterine device)
    * patients with positioning of hormone releasing intrauterine systems
    * patients with bilateral tubal occlusion
    * patients with vasectomized partner
    * patients who practice sexual abstinence
17. Any disorder, unwillingness or inability, which in the investigator's opinion, might jeopardise the subject's safety or compliance with the protocol
18. Previous surgical treatment for obesity (excluding liposuction >1 year before trial entry); 19 ) Inflammatory bowel diseases; 20 ) recent antibiotic therapy ( within 30 days before screening)

Cardiovascular- related

* Any of the following: myocardial infarction, stroke, hospitalisation for unstable angina pectoris or transient ischaemic attack within the past 60 days prior to the day of screening
* Planned coronary, carotid or peripheral artery revascularisation known on the day of screening;
* Presently classified as being in New York Heart Association (NYHA) Class IV heart failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-01-09 (Actual); Primary Completion 2020-01-09 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in gut microbiome composition assessed by Firmicutes-to-Bacteroidetes ratio using Quantitative polymerase chain reaction (PCR) | Change from baseline in gut microbiome composition at weeks 5 (visit 7)
  The liraglutide treatment effect on gut microbiome composition quantified as Firmicutes-to-Bacteroidetes ratio by Quantitative polymerase chain reaction (PCR)

SECONDARY OUTCOMES:
Change in body weight (kg) assessed by scale | Change from baseline in body weight at weeks 5 (visit 7)
  The liraglutide treatment effect on weight ( kg) assessed by scale
Change in body weight (kg) that will be combined with height (m) to report BMI (kg/m^2) where kg is a person's weight in kilograms and m2 is a person's height in metres squared | Change from baseline in body mass index at weeks 5 (visit 7)
  The liraglutide treatment effect on body weight (kg) that will be combined with height (m) to report BMI (kg/m^2) where kg is a person's weight in kilograms and m2 is a person's height in metres squared
Change in body composition assessed by Bioelectrical impedance analysis (BIA) | Change from baseline in body composition at weeks 5 (visit 7)
  The liraglutide treatment effect on body composition assessed by BIA
Change in hormonal regulation of appetite assessed by ghrelin levels | Change from baseline in ghrelin levels at weeks 5 (visit 7)
  The liraglutide treatment effect on hormonal regulation of appetite assessed by ghrelin levels
Change in hormonal regulation of hunger suppression assessed by cholecystokinin levels | Change from baseline in cholecystokinin levels at weeks 5 (visit 7)
  The liraglutide treatment effect on hormonal regulation of hunger suppression assessed by cholecystokinin levels
Change in hormonal regulation of appetite assessed by polipeptide YY levels | Change from baseline in polipeptide YY levels at weeks 5 (visit 7)
  The liraglutide treatment effect on hormonal regulation of appetite assessed by polipeptide YY levels
Change in hormonal regulation of weight assessed by leptin levels | Change from baseline in leptin levels at weeks 5 (visit 7)
  The liraglutide treatment effect on hormonal regulation of weight assessed by leptin levels
Change in low grade inflammation assessed by C-reactive protein levels | Change from baseline in C-reactive protein levels at weeks 5 (visit 7)
  The liraglutide treatment effect on low grade inflammation assessed by C-reactive protein levels
Change in low grade inflammation assessed by erythrocyte sedimentation rate (ESR) levels | Change from baseline in ESR levels at weeks 5 (visit 7)
  The liraglutide treatment effect on low grade inflammation assessed by ESR levels
Change in low grade inflammation assessed by interleukin- 1 (IL- 1) levels | Change from baseline in IL- 1 levels at weeks 5 (visit 7)
  The liraglutide treatment effect on low grade inflammation assessed by IL- 1 levels
Change in low grade inflammation assessed by interleukin- 6 (IL- 6) levels | Change from baseline in IL- 6 levels at weeks 5 (visit 7)
  The liraglutide treatment effect on low grade inflammation assessed by IL- 6 levels
Change in low grade inflammation assessed by interleukin- 10 (IL- 10) levels | Change from baseline in IL- 10 levels at weeks 5 (visit 7)
  The liraglutide treatment effect on low grade inflammation assessed by IL- 10 levels
Change in low grade inflammation assessed by Tumor Necrosis Factor -α (TNF-α) levels | Change from baseline in TNF-α levels at weeks 5 (visit 7)
  The liraglutide treatment effect on low grade inflammation assessed by TNF-α levels
Change in low grade inflammation assessed by monocyte chemotactic protein - 1 (MCP-1) levels | Change from baseline in MCP-1 levels at weeks 5 (visit 7)
  The liraglutide treatment effect on low grade inflammation assessed by MCP-1 levels
Change in lipid profile assessed by total cholesterol levels | Change from baseline in total cholesterol levels at weeks 5 (visit 7)
  The liraglutide treatment effect on lipid profile assessed by total cholesterol levels
Change in lipid profile assessed by LDL cholesterol levels | Change from baseline in LDL cholesterol levels at weeks 5 (visit 7)
  The liraglutide treatment effect on lipid profile assessed by LDL cholesterol levels
Change in lipid profile assessed by HDL cholesterol levels | Change from baseline in HDL cholesterol levels at weeks 5 (visit 7)
  The liraglutide treatment effect on lipid profile assessed by HDL cholesterol levels
Change in lipid profile assessed by triglycerides levels | Change from baseline in triglycerides levels at weeks 5 (visit 7)
  The liraglutide treatment effect on lipid profile assessed by triglycerides levels
Change in insulin resistance assessed by Matsuda Index | Change from baseline in insulin resistance assessed by Matsuda Index at weeks 5 (visit 7)
  The liraglutide treatment effect on insulin resistance assessed by Matsuda Index
Change in insulin resistance assessed by homeostasis model assessment - insulin resistance (HOMA-IR) Index | Change from baseline in insulin resistance assessed by HOMA-IR Index at weeks 5 (visit 7)
  The liraglutide treatment effect on insulin resistance assessed by HOMA-IR Index

CONTACTS AND LOCATIONS:
Locations (1):
- "Federico II" University of Naples, Department of Clinical and Molecular Endocrinology and Oncology, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eckburg PB, Bik EM, Bernstein CN, Purdom E, Dethlefsen L, Sargent M, Gill SR, Nelson KE, Relman DA. Diversity of the human intestinal microbial flora. Science. 2005 Jun 10;308(5728):1635-8. doi: 10.1126/science.1110591. Epub 2005 Apr 14. PMID 15831718
- [Background] Patterson E, Ryan PM, Cryan JF, Dinan TG, Ross RP, Fitzgerald GF, Stanton C. Gut microbiota, obesity and diabetes. Postgrad Med J. 2016 May;92(1087):286-300. doi: 10.1136/postgradmedj-2015-133285. Epub 2016 Feb 24. PMID 26912499
- [Background] Dinan TG, Cryan JF. Mood by microbe: towards clinical translation. Genome Med. 2016 Apr 6;8(1):36. doi: 10.1186/s13073-016-0292-1. PMID 27048547
- [Background] Nakatani Y, Maeda M, Matsumura M, Shimizu R, Banba N, Aso Y, Yasu T, Harasawa H. Effect of GLP-1 receptor agonist on gastrointestinal tract motility and residue rates as evaluated by capsule endoscopy. Diabetes Metab. 2017 Oct;43(5):430-437. doi: 10.1016/j.diabet.2017.05.009. Epub 2017 Jun 23. PMID 28648835
- [Background] Backhed F, Ding H, Wang T, Hooper LV, Koh GY, Nagy A, Semenkovich CF, Gordon JI. The gut microbiota as an environmental factor that regulates fat storage. Proc Natl Acad Sci U S A. 2004 Nov 2;101(44):15718-23. doi: 10.1073/pnas.0407076101. Epub 2004 Oct 25. PMID 15505215